CLINICAL TRIAL: NCT03267134
Title: The Hydrus Microstent for Refractory Open-Angle Glaucoma: A Prospective, Multicenter Clinical Trial (Hydrus VII Study)
Brief Title: Hydrus Microstent for Refractory Open-Angle Glaucoma
Acronym: SUMMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivantis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 16-001
Record Dates: First submitted 2017-08-22; First posted 2017-08-30 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Open-angle Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Ophthalmologic Surgical Procedures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hydrus Microstent (Experimental): Hydrus Microstent implanted in the eye per the supplied Hydrus Microstent Instructions for Use and associated training. Only one eye (study eye) will be implanted.
  Interventions: Device: Hydrus Microstent; Procedure: Ophthalmic surgery

INTERVENTIONS:
Device: Hydrus Microstent — Device implanted into the Schlemm's canal of the eye to provide a natural outflow pathway for aqueous humor, leading to a reduction in intraocular pressure (IOP). The Hydrus Microstent is intended for lifetime use of the glaucoma patient.
Procedure: Ophthalmic surgery — Implantation of the Hydrus Microstent performed under either local or topical ophthalmic anesthesia

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of the Hydrus Microstent in patients with refractory open-angle glaucoma.

DETAILED DESCRIPTION:
Participants will attend a screening visit, a baseline visit, a surgery visit, and 8 post-operative visits (Day 1, Day 7, Month 1, Month 2, Month 3, Month 6, Month 9, Month 12), for a total individual duration of approximately 14 months.

ELIGIBILITY:
Inclusion Criteria:

* Open-angle glaucoma with optic nerve pathology;
* BCVA of 20/80 or better in study eye;
* Refractory glaucoma;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Secondary glaucoma other than pseudoexfoliative and pigmentary glaucoma;
* Acute angle closure, chronic angle closure, or congenial, malignant, or developmental glaucoma;
* Pre-perimetric glaucoma;
* Ocular hypertension
* Shallow or flat anterior chamber;
* Other protocol-specified exclusion criteria may apply.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Lead, CRD Surgical, Study Director — Alcon Research, LLC
Locations (20):
- United States (16):
  - Vold Vision, Fayetteville, Arkansas
  - Sacramento Eye Consultants, Sacramento, California
  - Eye Center of Northern Colorado, Fort Collins, Colorado
  - Ocala Eye, Ocala, Florida
  - Center for Sight, Venice, Florida
  - Stiles Eyecare, Overland Park, Kansas
  - Louisiana Eye and Laser Center, Alexandria, Louisiana
  - Washington University in St. Louis Ophthalmology, St Louis, Missouri
  - Scott & Christie and Associates, Cranberry Township, Pennsylvania
  - Texan Eye, Austin, Texas
  - Glaucoma Associates of Texas, Dallas, Texas
  - El Paso Eye Surgeons, El Paso, Texas
  - Ophthalmology Associates, Fort Worth, Texas
  - Vale-Asche Russell Clinical Research Center, Houston, Texas
  - R and R Research, LLC, San Antonio, Texas
  - The Eye Centers of Racine and Kenosha, Kenosha, Wisconsin
- Clínica Oftalmológica, Barranquilla, Colombia
- Asian Eye Institute, Makati City, Philippines
- Hospital Universitario Miguel Servet, Zaragoza, Spain
- Manchester Royal Eye Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 20 investigative sites located in the United States (16), Philippines (1), Spain (1), United Kingdom (1), and Colombia (1).
Pre-assignment Details: Of the 217 subjects who signed an informed consent, 117 were exited from the study prior to attempted implantation as screen failures. This reporting group includes all subjects for whom a Hydrus Microstent was implanted or implantation was attempted (100) (Safety Analysis Population).
Units Other Than Participants: eyes
Groups:
- Hydrus Microstent: Hydrus Microstent implanted in the eye per the supplied Hydrus Microstent Instructions for Use and associated training, Only one eye (study eye) was implanted.
Period: Overall Study
Arm/Group | Hydrus Microstent
Started | 100; 100 eyes
Completed | 100; 100 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Safety Analysis Population
Arm/Group | Hydrus Microstent
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (10.0)
Age, Customized [Number; unit: participants]
  Less than 60 years | 13
  60 years to less than 70 years | 28
  70 to less than 80 years | 35
  80 years and greater | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 7
  Black or African American | 14
  Mestizo | 2
  White | 74
  Refuses to Answer/Unknown | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Greater Than or Equal to a 20 Percent Decrease From Baseline in Mean Diurnal Intraocular Pressure (MDIOP) at Month 12 While Maintaining the Same or Fewer Number of Medications as at Baseline
Description: Intraocular pressure was measured using Goldmann Applanation tonometry. Three separate IOP measurements were taken over an 8-hour period and averaged together to achieve mean diurnal intraocular pressure.
Time Frame: Baseline, Month 12
Population: Effectiveness Population: All subjects who undergo the Hydrus implantation surgery and are not discontinued early from the study due to unrelated reasons such as death or relocation. For non-responders, data was imputed as specified in the protocol. No hypothesis testing was pre-specified for this outcome measure.
Measure: Number; unit: percentage of subjects
Arm/Group | Hydrus Microstent
Number analyzed (Participants) | 100
percentage of subjects | 43.0

2. Secondary Outcome: Mean Change From Baseline in MDIOP at Month 12
Description: Intraocular pressure was measured using Goldmann Applanation tonometry and recorded in millimeters mercury (mmHG). Three separate IOP measurements were taken over an 8-hour period and averaged together to achieve mean diurnal intraocular pressure. A negative number represents a reduction from baseline. For non-responders, data was imputed as specified in the protocol. No hypothesis testing was pre-specified for this outcome measure.
Time Frame: Baseline, Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHG
Units Other Than Participants: eyes
Arm/Group | Hydrus Microstent
Number analyzed (Participants) | 100
Number analyzed (eyes) | 100
mmHG | -3.77 (5.0)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the operative visit to study exit (approximately 12 months). AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator.
Description: An adverse event (AE) was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the Microstent or delivery system.
Groups:
- Ocular Adverse Events; Non-Ocular Adverse Events: Hydrus Microstent implanted in the eye per the supplied Hydrus Microstent Instructions for Use and associated training, Only one eye (study eye) was implanted.
Arm/Group | Ocular Adverse Events | Non-Ocular Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 5/100 | 0/100
Other Adverse Events (participants affected / at risk) | 55/100 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ocular Adverse Events (N=100) | Non-Ocular Adverse Events (N=100)
Elevated IOP (Eye disorders) | 1 | 0
Elevated mean IOP (Eye disorders) | 2 | 0 — Equal or greater than 10 mmHg from baseline, greater than 1 month postoperatively
Worsening of visual field (Eye disorders) | 3 | 0 — Mean deviation equal or greater than 3 dB confirmed by 2 repeat measurements
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ocular Adverse Events (N=100) | Non-Ocular Adverse Events (N=100)
AC cell or flare requiring change in steroid medication regimen (Eye disorders) | 6 | 0
BCVA loss at greater than 1 month postoperative (Eye disorders) | 15 | 0 — BCVA loss defined as greater than or equal to 2 lines from baseline (ETDRS)
BCVA loss at less than or equal to 1 month postoperative (Eye disorders) | 10 | 0 — BCVA loss defined as greater than or equal to 2 lines from baseline (ETDRS)
Device obstruction (Eye disorders) | 10 | 0
Elevated mean IOP at greater than 1 month postoperative (Eye disorders) | 14 | 0 — Elevated mean IOP defined as IOP increase equal or greater than 10 mmHg from baseline
Elevated mean IOP at less than or equal to 1 month postoperative (Eye disorders) | 16 | 0 — Elevated mean IOP defined as IOP increase equal or greater than 10 mmHg from baseline
Hypotony (less than 6 mmHg) (Eye disorders) | 7 | 0
Surgical re-intervention in study eye (Eye disorders) | 15 | 0 — Not paracentesis within the 1 week visit
Worsening of visual field (Eye disorders) | 19 | 0 — Mean deviation greater than or equal to 3 dB confirmed by 2 repeat measurements

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT03267134/Prot_SAP_001.pdf